CLINICAL TRIAL: NCT03673722
Title: A Randomised Controlled Trial Investigating the Feasibility of a Multi-domain Intervention to Increase Mediterranean Diet (MedDiet) Score and Physical Activity (PA) of Older UK Adults Who Are at Above Average Risk of Dementia
Brief Title: Mediterranean Diet, Exercise and Dementia Risk in UK Adults
Acronym: MedEx-UK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of East Anglia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ARUK-PRRF2017-006UK
Record Dates: First submitted 2018-08-17; First posted 2018-09-17 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2018-08

CONDITIONS: Dementia
Keywords: Mediterranean Diet; Physical Activity; Dementia; Alzheimer Disease; Cognition
MeSH Terms: conditions — Dementia; Motor Activity; Alzheimer Disease | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: RCT
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MDP only (Experimental): Participants will be asked to increase their consumption of foods that are consistent with a Mediterranean Dietary Pattern through interaction with the online LEAP2 platform
  Interventions: Other: Foods consistent with a MDP
- MDP plus PA (Experimental): Participants will be asked to increase their consumption of foods that are consistent with a Mediterranean Dietary Pattern AND to increase Physical Activity using a mixture of structured and non-structured activities through interaction with the online LEAP2 platform
  Interventions: Other: Foods consistent with a MDP; Other: Physical Activity
- Control (Placebo Comparator): Participants will be given generic healthy eating advice based on the NHS 'Eatwell' plate and British Heart Foundation (BHF) guidelines
  Interventions: Other: Control

INTERVENTIONS:
Other: Foods consistent with a MDP — We aim to increase MDP by 3 points, according to a 14-point MEDAS score
  Arms: MDP only; MDP plus PA
Other: Physical Activity — We aim to increase PA to 150 minutes moderate activity per week.
  Arms: MDP plus PA
Other: Control — Participants will be given generic healthy eating advice based
  Arms: Control

SUMMARY:
In cohort studies, a Mediterranean Dietary Pattern (MDP) has been consistently associated with reduced dementia incidence. The efficacy of a MDP to prevent dementia has never been directly demonstrated by RCTs, with existing research limited to cognition as a secondary outcome. Furthermore, despite their likely additive effects, the combined impact of Physical Activity (PA) and a MDP on dementia risk is unknown.

MedEx-UK is a RCT that will evaluate the feasibility of a multi-domain intervention to increase Mediterranean Dietary Pattern (MDP) adherence and physical activity (PA) in a group of older UK adults who are at above average risk of dementia.

DETAILED DESCRIPTION:
In MedEx-UK the investigators propose to conduct a feasibility study in three UK centres (Norwich, Birmingham, Newcastle) which collectively will recruit 108 UK older adults (55-74y) who are at above average risk of dementia, but pre-clinical. Primary outcome is to evaluate the feasibility of a multi-domain intervention to increase MDP adherence and PA over a 24 week period, and to demonstrate the possibility of achieving meaningful behavioural change in a UK population. Secondary outcomes will be to measure the sensitivity of various cognitive assessments and measure the variability of our primary and secondary outcome measures in this population at baseline and in response to intervention.

There are three intervention arms to the study, and participants will be randomised with minimisation for gender and Mediterranean Diet Adherence Screener score (MEDAS; a validated questionnaire)

1. MDP:

   Participants will be asked to alter their consumption of foods consistent with a Mediterranean Diet. Examples include increased intake of fruits and vegetables, nuts, olive oil as the main culinary fat, moderate wine consumption (if they already consume alcohol), preferring white meat over red, and a reduction in commercial sweet and pastries, and sugar-sweetened drinks.
2. MDP plus PA:

   As well as the dietary intervention as in 1., participants will be asked to increase their PA using a mixture of structured (e.g. dancing, Zumba classes, swimming etc.) and non-structured (walking up stairs, gardening etc.) activities.
3. Control:

Participants will be given generic healthy eating advice based on the NHS 'Eatwell' plate and UK British Heart Foundation (BHF) guidelines.

The overall purpose of this study is to inform the feasibility and design of a future large-scale UK dementia risk reduction RCT, to observe whether a multi-domain intervention over 2 to 5 years promoting MDP adherence and increased PA can reduce cognitive decline and brain atrophy in adults at above average risk of dementia.

ELIGIBILITY:
Inclusion Criteria:

* Male and female, aged 55-74 years
* Understands and is willing and able to comply with all study procedures, including changes to diet and physical activity levels
* Access to, and able to use, the internet/computer/tablet device
* QRISK3 score of >=15 (assessed by GP)
* Subjective Memory Complaints (SMC), based on a score of >16 on the Cognitive Change Index (CCI) (from the first 12 items)
* Stable use of any prescribed medication for at least four weeks
* Normal (or corrected to normal) vision and hearing
* Fluent in written and spoken English
* Willing and able to provide written informed consent

Exclusion Criteria:

* Diagnosis of Alzheimer's disease (AD), other form of dementia, Mild Cognitive Impairment (MCI), or significant neurological disorder
* Cognition not within normal range, based on a score of <26 on the Montreal Cognitive Assessment (MoCA); or an indication of cognitive decline, based on a score of ≥2 on Ascertain Dementia (AD-8)
* Evidence of impairment of Instrumental Activities of Daily living (IADLS)
* Moderate to severe depression, assessed by the Patient Health Questionnaire (PHQ-9), a score of >10 being exclusionary
* Moderate to severe anxiety, assessed by the Generalised Anxiety Disorder Assessment (GAD-7), a score of >10 being exclusionary
* Current psychotic illness (delusional disorder/schizophrenia)
* History of serious mental illness know to affect cognition (schizophrenia, schizoaffective disorder, bipolar disorder)
* Subjects with other clinically diagnosed psychiatric disorders likely to affect the cognitive measures (as judged by a clinical advisor)
* HIV positive
* Past history or previous MRI evidence of brain damage, significant head trauma (including loss of consciousness as a result), brain surgery, stroke, or serious neurological disorders
* History of alcohol or drug dependency in the last 2 years
* Subjects with existing diagnosed gastrointestinal disorders likely to impact study results (as judged by a clinical advisor)
* History of any major cardiovascular event, such as a myocardial infarction, stroke or TIA
* Diagnosed COPD
* Cancer, or cancer/treatment within the last 12 months
* Diagnosis of type 1 or type 2 diabetes < 3 months ago
* Clinical diagnosis of liver or kidney disease
* Diagnosed Epilepsy
* Subjects with any other existing medical conditions likely to affect the study measures
* BMI >40kg/m2
* A habitual Mediterranean Diet Score (MDS) ≥9
* Habitual physical activity of >60 minutes moderate activity per week, assessed using the International Physical Activity Questionnaire (IPAQ), short form
* Currently actively engaged in a weight loss, other dietary, or physical activity intervention
* Prescribed medications likely to influence the study measures (as judged by a clinical advisor)
* Currently a participant or have participated in any other study involving an investigational product in the last 4 weeks
* Metal implants, e.g. pacemaker that precludes MRI.
* Claustrophobic which precludes MRI scanning.

Ages: 55 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2021-02-26 (Actual); Study Completion 2023-09-07 (Actual)

PRIMARY OUTCOMES:
Increase in MDP using the 14-point MEDAS scale | 24 weeks
  The extent to which the Mediterranean Dietary Pattern has improved, the target being an increase in 3 points of a 14-point scale, as assessed by Dietary Recall software (Intake 24) and a validated questionnaire (14-point MEDAS)
Increase in PA using activity monitors | 24 weeks
  The extent to which Physical Activity levels have increased, the target being 150 minutes of moderate activity per week, assessed using an activity monitor worn by participants throughout the 24 week intervention period

SECONDARY OUTCOMES:
Cognition | 24 weeks
  Cognitive test performance using a neuropsychological test battery which assesses various measures of global and domain specific function
Neuroimaging | 24 weeks
  MRI to assess regional blood flow and changes in brain structure
Vascular function | 24 weeks
  Assessed using Flow Mediated Dilation
QRISK3 score | 24 weeks
  Using a measurement of participant cholesterol levels and other data needed to calculate QRISK3 score (which assesses CVD risk; see www.qrisk.org/three/)
Blood pressure | 24 weeks
  Measurements of brachial artery blood pressure and 24 hour Ambulatory Blood Pressure
Blood markers | 24 weeks
  Selected inflammatory cytokines, nitric oxide metabolites and brain derived neurotrophic factor (BDNF)
Process evaluation | After 24 weeks
  Using a structured questionnaire and focus groups

CONTACTS AND LOCATIONS:
Overall Officials: Anne Marie Minihane, PhD, Principal Investigator — University of East Anglia
Locations (3):
- United Kingdom (3):
  - University of Birmingham, Birmingham
  - Newcastle University, Newcastle upon Tyne
  - University of East Anglia, Norwich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jennings A, Shannon OM, Gillings R, Lee V, Elsworthy R, Bundy R, Rao G, Hanson S, Hardeman W, Paddick SM, Siervo M, Aldred S, Mathers JC, Hornberger M, Minihane AM. Effectiveness and feasibility of a theory-informed intervention to improve Mediterranean diet adherence, physical activity and cognition in older adults at risk of dementia: the MedEx-UK randomised controlled trial. BMC Med. 2024 Dec 23;22(1):600. doi: 10.1186/s12916-024-03815-z. PMID 39716203
- [Derived] Elsworthy RJ, Jong ST, Hanson S, Shannon OM, Jennings A, Gillings R, Siervo M, Hornberger M, Hardeman W, Mathers JC, Minihane AM, Aldred S. Effects of the COVID-19 associated United Kingdom lockdown on physical activity in older adults at high risk of cardiovascular disease: a mixed methods perspective from the MedEx-UK multicenter trial. Front Public Health. 2024 May 9;12:1371453. doi: 10.3389/fpubh.2024.1371453. eCollection 2024. PMID 38784572
- [Derived] Shannon OM, Lee V, Bundy R, Gillings R, Jennings A, Stephan B, Hornberger M, Balanos G, Paddick SM, Hanson S, Hardeman W, Holmes R, Garner N, Aldred S, Siervo M, Mathers JC, Minihane AM. Feasibility and acceptability of a multi-domain intervention to increase Mediterranean diet adherence and physical activity in older UK adults at risk of dementia: protocol for the MedEx-UK randomised controlled trial. BMJ Open. 2021 Feb 5;11(2):e042823. doi: 10.1136/bmjopen-2020-042823. PMID 33550254